CLINICAL TRIAL: NCT01738711
Title: Does Cognitive Behavioural Therapy (CBT) Delivered by a Respiratory Nurse Reduce Anxiety and the Impact of Cough and Breathlessness on Quality of Life in Patients With Idiopathic Pulmonary Fibrosis (IPF)?
Brief Title: Does CBT Improve the Perception/Impact of Cough and Breathlessness in IPF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Victoria Infirmary (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Ian Forrest, Consultant Respiratory Physician, Royal Victoria Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPF Protocol 12/NE/0309
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cough; Breathlessness
Keywords: Idiopathic pulmonary fibrosis; Cognitive behavioural therapy; Anxiety; Quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough; Dyspnea; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioural Therapy (Active Comparator): Patient in this arm receive 2-6 sessions of cognitive behavioural therapy
  Interventions: Behavioral: Cognitive behavioural therapy
- Written information on CBT (Placebo Comparator): Patients in this arm do not receive sessions of CBT but receive written information on anxiety control as per standard practice

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — Patient receive 2-6 sessions depending on individual need. first session is 1 hour duration with additional sessions approximately 30 minutes.
  Other Names: CBT
  Arms: Cognitive Behavioural Therapy

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic progressive lung disease of unknown cause for which there is no effective medical treatment. The main symptoms are increasing breathlessness and cough which can significantly impact on quality of life (QOL) often leading to anxiety and depression. The focus of disease management is shifting from pharmacological attempts to reduce disease progression to managing symptoms and a more holistic approach. Cognitive behavioural therapy (CBT) is increasingly used to treat anxiety and depression in chronic disease. Our investigators aim to determine whether CBT can reduce anxiety and depression related to symptoms and improve QOL in patients with IPF. This study will compare CBT intervention (Group 1) against standard treatment (Group 2). Patients will be recruited from a specialist IPF clinic - all patients attending with IPF who suffer from anxiety will be eligible to participate in the study. The study aims to recruit 30 patients (15 in each group). Patients will be randomly allocated into each group using an envelope concealment system. At entry a baseline visit will be conducted with information gathered regarding disease severity, hospital admissions, medication, symptoms (subjective and objective), quality of life and anxiety and depression using questionnaires and routine clinical tests. Patients will then receive CBT intervention (Group 1) or no intervention (Group 2). Patients receiving CBT will undergo a maximum of 6 (minimum of 2) individual therapy sessions. Follow up visits for both groups will be conducted at 3, 6, 9 and 12 months with the same information gathered as at the baseline visit.

DETAILED DESCRIPTION:
Medical therapies (e.g. prednisolone, azathioprine and N-acetylcysteine) have not shown any benefit in patients with IPF and may cause harm. Therefore the focus of management has shifted towards a more holistic approach-management of the symptoms and how patients cope with these, in a chronic progressive terminal disease. Anxiety is recognised to contribute to patients' perceptions of symptoms and quality of life. CBT is being increasingly used in other chronic respiratory diseases, such as chronic obstructive pulmonary disease (COPD) where there is some evidence that it reduces anxiety and breathlessness. Currently there is no evidence regarding its use in IPF. If CBT is shown to reduce anxiety and help patients cope with symptoms of cough and breathlessness then it can be integrated into the care of all IPF patients to improve quality of life.

All patients attending our specialist IPF clinic will be asked to complete a hospital anxiety and depression questionnaire (HADS). All those with anxiety (HADS-A of equal to or greater than 8) will be eligible for entry. Study information will be provided to these patients and they will then be contacted between 24 and 48 hours later by telephone to confirm they wish to enter the study. If they wish to participate a hospital visit will be arranged to complete informed consent, gather baseline information and be randomised. If allocated to the CBT intervention group they will then receive a maximum of 6 (minimum of 2) sessions of CBT on an individual basis. Patients allocated to the placebo group will receive written information on anxiety management. All patients will attend four more clinic visits at three, six, nine and twelve months after randomisation. At each clinic visit they will complete five questionnaires (totalling 60 questions) and undergo lung function and six minute walk test. They will be consented to wear a cough monitor for a 24 hour period at both baseline and 3 month visits. The cough monitor records the number of times a patient coughs and how long they cough for during a 24 hour period. A small microphone is attached to the clothing and another small microphone to the chest wall which is connected to a small recording device. The device is carried around the waist. The patient will then return the cough monitor the following day. The monitor records not only coughing sounds but also other sounds around the microphone. However, computer software is used to remove parts of the recording where there is no sound, such as when reading or sleeping. It is also designed to remove distant noises, such as another person's conversation or noise from a television but this depends on how loud or close the noise is to the microphone.

The anonymised recordings will be analysed by a trained researcher at Manchester University who counts the number of coughs. The recordings are kept confidential and are stored anonymously at the University of Manchester for a period of 15 years.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of IPF confirmed by a specialist IPF MDT according to ATS/ERS criteria, agreement to participate and provide written, informed consent, agreement to attend a minimum of 2 and maximum of 6 CBT sessions.

Exclusion Criteria:

HADS-A equal or more than eight, Known psychiatric disorders, psychosis or personality disorders, currently receiving psychological therapy including counselling and/or cognitive behavioural therapy (CBT), cognitive impairment e.g. dementia preventing engagement with CBT, unwilling to engage in CBT, verbal and/or written communication problems limiting ability to engage with CBT or provide written consent (all attempts made to include patients in whom English is not their first language by using an interpreter).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
validity of tools used | baseline and 12 months
  to determine validity of tools used in pilot study to inform a future, multicentre RCT.
estimation of recruitment rate | baseline to 12 months
  to determine estimation of recruitment rate to inform a future RCT
number of patients needed | baseline to 12 months
  estimation of parameters such as variance of outcome variables to enable calculation of sample size in a future RCT.

SECONDARY OUTCOMES:
change in Hospital Anxiety and Depression Scale-Anxiety subset | baseline and 3 months
  to assess change in anxiety scores using the Hospital Anxiety and Depression Scale (anxiety subset) at 3 months.
change in Hospital Anxiety and Depression Scale-Depression subset | baseline and 3 months
  to assess change in depression using the Hospital Anxiety and Depression Scale (depression subset) at 3 months.
change in cough frequency | baseline and 3 months
  to assess change in cough frequency using a 24 hour cough monitor
change in Medical Research Council (MRC) dyspnoea scale | baseline and 3 months
  to assess the impact on breathlessness using change in MRC dyspnoea scale at 3 months
change in pulmonary function tests (FVC, TLCO) | baseline and 3 months
  to assess impact on disease severity using pulmonary function tests at 3 months
change in leicester cough questionnaire | baseline and 3 months
  to assess the change in quality of life using the Leicester cough questionnaire at 3 months
change in Hospital Anxiety and Depression Scale-Anxiety subset | baseline and 6 months
  change in anxiety score using Hospital Anxiety and Depression Scale (anxiety subset) at 6 months
change in Hospital Anxiety and Depression Scale-Anxiety subset | baseline and 9 months
  change in anxiety score using the Hospital Anxiety and Depression Scale (anxiety subset) at 9 months
change in Hospital Anxiety and Depression Scale-Anxiety subset | baseline and 12 months
  change in anxiety score using the Hospital Anxiety and Depression Scale (anxiety subset) at 12 months
change in Hospital Anxiety and Depression Scale-Depression subset | baseline and 6 months
  to assess change in depression using the Hospital Anxiety and Depression Scale (depression subset) at 6 months.
change in Hospital Anxiety and Depression Scale-Depression subset | baseline and 9 months
  to assess change in depression using the Hospital Anxiety and Depression Scale (depression subset) at 9 months.
change in Hospital Anxiety and Depression Scale-Depression subset | baseline and 12 months
  to assess change in depression using the Hospital Anxiety and Depression Scale (depression subset) at 12 months.
change in MRC dyspnoea scale | baseline and 6 months
  to assess the impact on breathlessness using change in MRC dyspnoea scale at 6 months
change in MRC dyspnoea scale | baseline and 9 months
  to assess the impact on breathlessness using change in MRC dyspnoea scale at 9 months
change in MRC dyspnoea scale | baseline and 12 months
  to assess the impact on breathlessness using change in MRC dyspnoea scale at 12 months
change in pulmonary function tests (FVC, TLCO) | baseline and 6 months
  to assess impact on disease severity using pulmonary function tests at 6 months
change in pulmonary function tests (FVC, TLCO) | baseline and 9 months
  to assess impact on disease severity using pulmonary function tests at 9 months
change in pulmonary function tests (FVC, TLCO) | baseline and 12 months
  to assess impact on disease severity using pulmonary function tests at 12 months
change in 6 minute walk distance | baseline and 3 months
  to assess impact on disease severity using six minute walk distance and desaturation index at 3 months
change in six minute walk distance | baseline and 6 months
  to assess impact on disease severity using six minute walk distance and desaturation index at 6 months
change in six minute walk distance | baseline and 9 months
  to assess impact on disease severity using six minute walk distance and desaturation index at 9 months
change in six minute walk distance | baseline and 12 months
  to assess impact on disease severity using six minute walk distance and desaturation index at 12 months
change in leicester cough questionnaire | baseline and 6 months
  to assess the change in quality of life using the Leicester cough questionnaire at 6 months
change in leicester cough questionnaire | baseline and 9 months
  to assess the change in quality of life using the Leicester cough questionnaire at 9 months
change in leicester cough questionnaire | baseline and 12 months
  to assess the change in quality of life using the Leicester cough questionnaire at 12 months
change in King's brief interstitial lung disease questionnaire | baseline and 3 months
  to assess the change in quality of life using the King's brief Interstitial Lung Disease questionnaire at 3 months
change in King's brief interstitial lung disease questionnaire | baseline and 6 months
  to assess the change in quality of life using the King's brief Interstitial Lung Disease questionnaire at 6 months
change in King's brief interstitial lung disease questionnaire | baseline and 9 months
  to assess the change in quality of life using the King's brief Interstitial Lung Disease questionnaire at 9 months
change in King's brief interstitial lung disease questionnaire | baseline and 12 months
  to assess the change in quality of life using the King's brief Interstitial Lung Disease questionnaire at 12 months
change in generalised anxiety disorder questionnaire | baseline and 3 months
  to assess the change in quality of life using the Generalised anxiety disorder questionnaire at 3 months
change in generalised anxiety disorder questionnaire | baseline and 6 months
  to assess the change in quality of life using the Generalised anxiety disorder questionnaire at 6 months
change in generalised anxiety disorder questionnaire | baseline and 9 months
  to assess the change in quality of life using the Generalised anxiety disorder questionnaire at 9 months
change in generalised anxiety disorder questionnaire | baseline and 12 months
  to assess the change in quality of life using the Generalised anxiety disorder questionnaire at 12 months
change in EuroQol5 Dimension questionnaire | baseline and 3 months
  to assess the change in quality of life using the EuroQol5 Dimension questionnaire at 3 months
change in EuroQol5 Dimension questionnaire | baseline and 6 months
  to assess the change in quality of life using the EuroQol5 Dimension questionnaire at 6 months
change in EuroQol5 Dimension questionnaire | baseline and 9 months
  to assess the change in quality of life using the EuroQol5 Dimension questionnaire at 9 months
change in EuroQol5 Dimension questionnaire | baseline and 12 months
  to assess the change in quality of life using the EuroQol5 Dimension questionnaire at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian Forrest, MRCP UK, PhD, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom, United Kingdom

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Brown KK. Chronic cough due to chronic interstitial pulmonary diseases: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):180S-185S. doi: 10.1378/chest.129.1_suppl.180S. PMID 16428708
- [Background] de Godoy DV, de Godoy RF. A randomized controlled trial of the effect of psychotherapy on anxiety and depression in chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2003 Aug;84(8):1154-7. doi: 10.1016/s0003-9993(03)00239-9. PMID 12917854
- [Background] Doherty MJ, Mister R, Pearson MG, Calverley PM. Capsaicin induced cough in cryptogenic fibrosing alveolitis. Thorax. 2000 Dec;55(12):1028-32. doi: 10.1136/thorax.55.12.1028. PMID 11083888
- [Background] Eiser N, West C, Evans S, Jeffers A, Quirk F. Effects of psychotherapy in moderately severe COPD: a pilot study. Eur Respir J. 1997 Jul;10(7):1581-4. doi: 10.1183/09031936.97.10071581. PMID 9230251
- [Background] Heslop K, De Soyza A, Baker CR, Stenton C, Burns GP. Using individualised cognitive behavioural therapy as a treatment for people with COPD. Nurs Times. 2009 Apr 14-20;105(14):14-7. PMID 19449602
- [Background] Hope-Gill BD, Hilldrup S, Davies C, Newton RP, Harrison NK. A study of the cough reflex in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2003 Oct 15;168(8):995-1002. doi: 10.1164/rccm.200304-597OC. Epub 2003 Aug 13. PMID 12917229
- [Background] Jones RM, Hilldrup S, Hope-Gill BD, Eccles R, Harrison NK. Mechanical induction of cough in Idiopathic Pulmonary Fibrosis. Cough. 2011 Apr 10;7:2. doi: 10.1186/1745-9974-7-2. PMID 21477349
- [Background] Madison JM, Irwin RS. Chronic cough in adults with interstitial lung disease. Curr Opin Pulm Med. 2005 Sep;11(5):412-6. doi: 10.1097/01.mcp.0000174249.07762.37. PMID 16093815
- [Background] Patel AS et al. The assessment of health related quality of life in interstitial lung disease with the King's brief interstitial lung disease questionnaire (K-ILD). Thorax 2011: A61
- [Background] Ryerson CJ, Collard HR, Pantilat SZ. Management of dyspnea in interstitial lung disease. Curr Opin Support Palliat Care. 2010 Jun;4(2):69-75. doi: 10.1097/SPC.0b013e3283392b51. PMID 20375900
- [Background] Shipley MD, Hardy T, Heslop K, Forrest IA. Identifying anxiety and depression in interstitial lung disease: use of a simple outpatient screening tool. British Thoracic Society Winter Meeting 2009
- [Background] Bradley B, Branley HM, Egan JJ, Greaves MS, Hansell DM, Harrison NK, Hirani N, Hubbard R, Lake F, Millar AB, Wallace WA, Wells AU, Whyte MK, Wilsher ML; British Thoracic Society Interstitial Lung Disease Guideline Group, British Thoracic Society Standards of Care Committee; Thoracic Society of Australia; New Zealand Thoracic Society; Irish Thoracic Society. Interstitial lung disease guideline: the British Thoracic Society in collaboration with the Thoracic Society of Australia and New Zealand and the Irish Thoracic Society. Thorax. 2008 Sep;63 Suppl 5:v1-58. doi: 10.1136/thx.2008.101691. No abstract available. PMID 18757459